CLINICAL TRIAL: NCT02436447
Title: A Phase 1, 7 Day Repeat Dose, Parallel-Group, Open-Label Study to Evaluate the Safety and Pharmacokinetics of Intravenous Infusion of MTP-131 Administered in Subjects With Impaired Renal Function
Brief Title: A Phase 1 Study Investigating the Safety and Pharmacokinetics of Repeat-dose Intravenous Infusion of MTP-131 in Subjects With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SPICP-101
Record Dates: First submitted 2015-04-30; First posted 2015-05-06 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Normal and Impaired Renal Function
Keywords: Renal Impairment, Renal function, MTP-131, Bendavia™
MeSH Terms: conditions — Renal Insufficiency | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal renal function (Experimental)
  Interventions: Drug: MTP-131
- Mild renal impairment (Experimental)
  Interventions: Drug: MTP-131
- Moderate renal impairment (Experimental)
  Interventions: Drug: MTP-131
- Severe renal impairment (Experimental)
  Interventions: Drug: MTP-131

INTERVENTIONS:
Drug: MTP-131 — MTP-131 administered as once-daily 1- hour intravenous infusion for 7 consecutive days in subjects with normal renal function.
  Arms: Normal renal function
Drug: MTP-131 — MTP-131 administered as once-daily 1- hour intravenous infusion for 7 consecutive days in subjects with mild renal impairment.
  Arms: Mild renal impairment
Drug: MTP-131 — MTP-131 administered as once-daily 1- hour intravenous infusion for 7 consecutive days in subjects with moderate renal impairment
  Arms: Moderate renal impairment
Drug: MTP-131 — MTP-131 administered as once-daily 1- hour intravenous infusion for 7 consecutive days in subjects with severe renal impairment
  Arms: Severe renal impairment

SUMMARY:
This study is a Phase 1, open-label, parallel group, multiple dose study, in subjects over 18 years, to evaluate the safety, tolerability, and pharmacokinetics of one-hour intravenous infusion of MTP-131 administered for 7 consecutive days. Twenty-four subjects are planned to be enrolled into 4 cohorts of varying renal function, with each cohort consisting of 6 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years-of-age at the Screening Visit.
* Subject has signed an ICF before any study specific procedures are performed.
* Subjects selected for each cohort must satisfy the following creatinine clearance (CLCR) criteria (as determined by 24 hour urine collection and analysis):

  * Cohort 1 - Normal Renal Function, 24 hour CLCR ≥ 90 mL/min
  * Cohort 2 - Mild renal impairment, 24 hour CLCR ≥ 60-89 mL/min
  * Cohort 3 - Moderate renal impairment, 24 hour CLCR ≥ 30-59 mL/min
  * Cohort 4 - Severe renal impairment, 24 hour CLCR <30 not requiring dialysis
* Have a history of stable renal impairment as determined by standard estimated creatinine clearance methodology (at least 1 month within the same descriptive cohort) and be in a stable physical condition based on findings of medical history.
* Women of childbearing potential must agree to use 1 of the following methods of birth control from the date they sign the ICF until two months after the last dose of study drug:

  1. Abstinence, when it is in line with the preferred and usual lifestyle of the subject. Subject agrees to use an acceptable method of contraception should they become sexually active.
  2. Maintenance of a monogamous relationship with a male partner who has been surgically sterilized by vasectomy (the vasectomy procedure must have been conducted at least 60 days prior to the Screening Visit or confirmed via sperm analysis).
  3. Barrier method (e.g., condom or occlusive cap) with spermicidal foam/gel/film/cream AND either hormonal contraception (oral, implanted, or injectable) or an intrauterine device or system.

Exclusion Criteria:

* Subject has history of any concurrent medical condition which, in the opinion of the investigator, significantly increases the potential risks associated with administration of MTP-131 or any other aspect of study participation, with the exception of renal impairment.
* Female subjects who are pregnant, planning to become pregnant, or lactating.
* Subject has history of cancer (with the exception of non-melanoma skin cancer), unless the subject has documentation of completed curative treatment
* Subject has history of renal transplantation.
* Subject has active inflammatory renal disease.
* Subject has a history of histamine intolerance (e.g., a known deficiency of endogenous or exogenous histamine degradation).
* Subject is currently receiving treatment with chemotherapeutic agents or immunosuppressant agents.
* Subject has positive serology for HIV 1, HIV 2, HBsAg or HCV.
* Subject has donated or received blood or blood products within the past 30 days.
* Subject participated in a clinical study involving investigational product within 30 days prior to the planned date of study drug administration.
* Subject has a history of clinically significant hypersensitivity or allergy to any of the excipients contained in the study drug.
* Subject has a history of active alcoholism or drug addiction during the year before the Screening Visit.

  * Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Mean peak plasma concentration (Cmax) of MTP-131 (ng/ml) in each cohort | Assessed up to Day 14

SECONDARY OUTCOMES:
Incidence of Adverse Events | Assessed up to Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Maimi, Florida, United States